CLINICAL TRIAL: NCT06833489
Title: Transcriptomic Analysis to Put an End to Misdiagnosis in Patients With Rare Muscle Diseases
Acronym: ARNseq-Musc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM22_0420; 2024-A01079-38 (Other: RCB)
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Rare Genetic Muscle Diseases; Muscular Dystrophy, Duchenne; Muscular Dystrophy, Becker; Congenital Myopathy; Pompe Disease (Infantile-Onset)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Myotonia Congenita; Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequencing of RNAseq libraries (Experimental): There will be no visits from participants, so we will be using samples already in the Biological Resources Centre (CRB).
  RNA will be extracted from muscle biopsies taken as part of the treatment. RNAseq libraries will be sequenced by the Genomics and Bioinformatics Platform (GBiM) at Marseille Medical Genetics (MMG, U1251, AMU). Sequencing will be performed in paired-end (2*100 bp) on Illumina's Novaseq 6000 system (50 million clusters per sample, 100 M paired-end reads) and then analysed by bioinformatics.
  Interventions: Other: ARN extraction from muscle biopsies

INTERVENTIONS:
Other: ARN extraction from muscle biopsies — There will be no visits from participants, so we will be using samples already in the Biological Resources Centre (CRB).
  RNA will be extracted from muscle biopsies taken as part of the treatment. RNAseq libraries will be sequenced by the Genomics and Bioinformatics Platform (GBiM) at Marseille Medical Genetics (MMG, U1251, AMU). Sequencing will be performed in paired-end (2*100 bp) on Illumina's Novaseq 6000 system (50 million clusters per sample, 100 M paired-end reads) and then analysed by bioinformatics.

SUMMARY:
Since 2017, more than 250 analyses performed at the Molecular Genetics Laboratory of the Timone Enfant Hospital have yielded negative results in patients with rare genetic muscle diseases. The researchers hypothesise that some of these misdiagnosed patients carry pathogenic RNA (transcript) disrupting variants that were not identified by DNA sequencing. In fact, DNA sequencing analyses can be negative despite the presence of a pathogenic variant that disrupts RNA splicing or expression, causing a genetic disease. For this reason, RNA sequencing can provide a diagnosis in patients who have not been diagnosed by DNA sequencing, thus putting an end to diagnostic wandering. Thus, as a descriptive prevalence study, the objectives are first to determine the rate of positive diagnoses made by the RNAseq approach in patients with muscle diseases that have not yet been diagnosed, and then to identify the genomic characteristics of the pathogenic variants identified in patients by RNAseq analysis, in order to facilitate the identification of this type of variant in future patients.

50 patients will be included in this study during 2 years.

ELIGIBILITY:
Inclusion Criteria:

* patients with rare genetic muscle diseases who have benefited from high-throughput sequencing analysis (panel of 200 genes defined by the FILNEMUS Rare Neuromuscular Disease Network) carried out at the Molecular Genetics Laboratory, Medical Genetics Department, Timone Enfant Hospital since 2017.

This criterion is necessary to limit the analysis to patients with muscular diseases among all the patients analysed by the Molecular Genetics Laboratory.

* this genetic analysis did not identify pathogenic variants explaining the patient's phenotype This criterion is necessary in order to include only patients in diagnostic error.
* a muscle biopsy of the patient is available in the Biological Resources Centre (CRB) at the AP-HM.

Exclusion Criteria:

* Patients with no muscle biopsy available in the CRB.
* Patients with an established molecular diagnosis.
* Patients for whom RNA extraction from a muscle biopsy sample did not yield RNA of sufficient quality (INR >7) will be excluded from the study. A maximum of two extraction attempts will be performed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
rate of positive diagnoses using the RNAseq approach | From enrollment to the end of study at 24 months
  to determine the rate of positive diagnoses made using the RNAseq approach in patients with muscle diseases who have not yet been diagnosed. A patient is considered to be in diagnostic limbo if DNA sequencing of 200 genes responsible for muscle diseases has not identified pathogenic variants responsible for the patient's phenotype. Investigators are going to use transcriptomic analysis (RNA sequencing) in combination with innovative bioinformatics tools to identify variants with a deleterious effect at RNA level in patients with undiagnosed muscle diseases. This will make it possible to establish a molecular diagnosis and put an end to misdiagnosis in many patients.

SECONDARY OUTCOMES:
Identification of genomic characteristics | From enrollment to end of study at 24 months
  identify the genomic characteristics of pathogenic variants identified by the RNAseq approach. This analysis could potentially uncover certain characteristics that are specific to this type of variant, making it possible to suggest their presence in other undiagnosed patients in the future.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Timone, Marseille, France